CLINICAL TRIAL: NCT07319689
Title: Predictors of Myasthenia Gravis Outcome Following Thoracoscopic Thymectomy: Multicenter Comparative Study Between Thymomatous and Non-Thymomatous Patients
Brief Title: Predictors of Myasthenia Gravis Outcome Following Thoracoscopic Thymectomy: Comparative Study Between Thymomatous and Non-Thymomatous Patients
Status: Completed | Type: Observational
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mostafa Mohamed Elawady, Lecturer of Neuropsychiatry, Tanta University, Tanta, Egypt., Tanta University
Other Study IDs: 36264PR13103/10/25
Record Dates: First submitted 2025-12-20; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Predictor; Myasthenia Gravis; Thoracoscopic Thymectomy; Thymomatous; Non-Thymomatous
MeSH Terms: conditions — Myasthenia Gravis | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Thymomatous Myasthenia Gravis group: Thymomatous myasthenia gravis (patients with histologically confirmed thymoma).
  Interventions: Other: Data collection
- Non-thymomatous Myasthenia Gravis group: Non-thymomatous myasthenia gravis (patients with thymic hyperplasia or normal/ involuted thymus).
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — Data were obtained from patient files, operative notes, and electronic medical records.

SUMMARY:
This study aimed to assess and compare predictors of outcome in patients with thymomatous and non-thymomatous MG undergoing Thoracoscopic thymectomy.

DETAILED DESCRIPTION:
Myasthenia Gravis (MG) is a chronic autoimmune neuromuscular disorder characterized by fluctuating muscle weakness resulting from antibodies that target acetylcholine receptors or associated proteins at the neuromuscular junction.

Thoracoscopic thymectomy becomes more prominent than traditional transsternal thymectomy due to fewer perioperative complications with shorter hospital stays and more favorable long-term outcomes.

Prognostic outcomes following thoracoscopic thymectomy can vary significantly between non-thymomatous and thymomatous MG, necessitating a thorough investigation of these differences.

ELIGIBILITY:
Inclusion Criteria:

* Both sexes.
* Confirmed diagnosis of Myasthenia Gravis (MG).
* Underwent Thoracoscopic thymectomy.
* Availability of complete preoperative and postoperative records, including imaging and histopathology.
* Minimum follow-up of 9 months post-surgery.

Exclusion Criteria:

* Patients who underwent thymectomy for indications other than MG.
* Incomplete medical records or loss to follow-up before outcome assessment.
* Patients with concomitant neuromuscular disorders other than MG

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study was a combined prospective and retrospective, observational, and comparative study conducted in the neurology and cardiothoracic departments at Tanta and Zagazig University Hospitals between January 2022 and December 2025.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2025-12-18 (Actual); Study Completion 2025-12-18 (Actual)

PRIMARY OUTCOMES:
Proportion of patients achieving complete stable remission | 12 months post-procedure
  Proportion of patients achieving complete stable remission was recorded.

SECONDARY OUTCOMES:
Proportion of patients achieving pharmacologic remission | 12 months post-procedure
  Proportion of patients achieving pharmacologic remission was recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.